CLINICAL TRIAL: NCT06753383
Title: Effectiveness of Virtual Reality- Based Rehabilitation Program in Individuals With Adolescent Idiopathic Scoliosis After Posterior Fusion Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Elif Yagmur Ozger (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Elif Yagmur Ozger, Sponsor-Investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/2091
Record Dates: First submitted 2024-12-16; First posted 2024-12-31 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: Adolescent Idiopathic Scoliosis; virtual reality based rehabilitation; Respiratory Muscle Strength; Posterior Fusion Surgery; spinal mobility; kinesiophobia; spinopelvic parameter
MeSH Terms: conditions — Kinesiophobia | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Based Exercise Group (Experimental): The Virtual Reality Based Exercise Group will be given an exercise program based on the games in Kinect Sports Ultimate (Soccer, Basketball, Skiing, Tennis, Baseball, Volleyball, Boxing, Track & Field) for 30 minutes a day for a total of 6 weeks, 2 days a week. The games include movements such as lateral flexion, extension and flexion of the torso and upper limb movements, running, short-urea standing on one leg, jumping.
  Interventions: Other: To the Virtual Reality Based Exercise
- Control Group (Active Comparator): The participants who make up the control group will be followed up with a routine physiotherapy and rehabilitation program for 6 weeks.
  Interventions: Other: Routine physiotherapy and rehabilitation program

INTERVENTIONS:
Other: To the Virtual Reality Based Exercise — After posterior fusion surgery, a rehabilitation program will be applied to individuals with AIS using Kinect Sports Ultimate for 30 minutes per day for a total of 6 weeks, 2 days a week.
  Arms: Virtual Reality Based Exercise Group
Other: Routine physiotherapy and rehabilitation program — 14 patients with posterior fusion AIS routinely in the postoperative clinic for 6 weeks. the physiotherapy program used will be applied.
  Arms: Control Group

SUMMARY:
The aim of this clinical study is to investigate the effect of virtual reality based rehabilitation program on kinesiophobia, respiratory muscle strength, spinal mobility, physical activity, spinopelvic parameters and quality of life after posterior fusion surgery in individuals diagnosed with Adolescent Idiopathic Scoliosis (AIS). The main questions it aims to answer are:

* Does a virtual reality based rehabilitation program after posterior fusion surgery have an effect on kinesiophobia, respiratory muscle strength, spinal mobility, physical activity, spinopelvic parameters and quality of life in individuals diagnosed with AIS?
* Is the virtual reality-based rehabilitation program after posterior fusion surgery more effective for individuals diagnosed with AIS than the routine physiotherapy and rehabilitation program applied in the clinic?

They will compare it with the [routine physiotherapy and rehabilitation program] to see if the virtual reality-based rehabilitation program is effective in individuals with AIS after posterior fusion.

Participants :

After being evaluated in terms of kinesiophobia, respiratory muscle strength, spinal mobility, physical activity, spinopelvic parameters and quality of life, the Virtual Reality-Based Exercise Group will be given an exercise program via the games in Kinect Sports Ultimate for 30 minutes a day for a total of 6 weeks, 2 days . At the end of the 6 week, the participants will be re-evaluated and the results will be compared according to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AIS December 10-18
* Underwent posterior spinal fusion surgery
* Post-operative (post-op) 6.during the week and after
* Absence of vision, speech and hearing problems
* Regular participation in the program to be implemented
* Volunteering of individuals

Exclusion Criteria:

* Have a history of previous spinal surgery
* Have any contraindications to exercise
* Have a mental problem
* Have a neuromuscular, mesenchymal, rheumatic disease
* Have pulmonary and cardiac complications

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-07-21 (Estimated)

PRIMARY OUTCOMES:
Spinal Mobility | 6 weeks
  The spinal mobility of the participants will be measured with the modified Schober test before and after 6 weeks of treatment. When the person is in an upright position, the lumbosacral junction and 10 cm above will be marked, and a third marker will be placed 5 cm below the lumbosacral junction. After the anterior flexion, which is performed as far forward as possible, the distance between the top and bottom deceleration will be measured and the test will be terminated.
Respiratory Muscle Strength | 6 weeks
  The respiratory muscle strength of the participants will be measured according to the criteria of the American Thoracic Society /European Respiratory Society using a portable, electronic intraoral pressure measuring device. After the maximum expiration, the participant will be asked to perform maximal inspiration lasting at least 1.5 seconds in the residual volume. At the total lung capacity after maximum inspiration, the person will be asked to perform a maximum expiration lasting at least 1.5 seconds against the closed system. The tests will be applied in a sitting position with the nose closed with a soft latch. Of at least three measurements that are technically acceptable and do not differ by more than 5 cmH₂O from each other, the highest one will be recorded.

SECONDARY OUTCOMES:
Spinopelvic Parameters | 6 weeks
  All the spinal anterior, posterior and lateral spine ortho x-rays of the participants and spinal parameters and pelvic parameters will be measured before and after virtual reality based rehabilitation applications and the effect of virtual reality based rehabilitation program on the sagittal balance of the spine will be examined
Physical Activity | 6 weeks
  Individuals with AIS will be taught to use pedometers and will be asked to use the device from the moment they get up in the morning until the moment they go to bed at night for 6 weeks, to record the number of steps values before going to bed at night.
Kinesiophobia | 6 weeks
  Participants' fear of movement will be questioned using the TAMPA Kinesiophobia scale. The minimum score that can be taken from the scale is 17 and the maximum score is 68. High scores indicate that the patient's fear of movement is high.
Scoliosis Quality of Life | 6 weeks
  The Scoliosis Research Society-22 Questionnaire (SRS-22) will be used to evaluate the health-related quality of life of individuals with AIS before and after rehabilitation practices performed via virtual reality. The score range for each item ranges from zero (worst) to five (best). Decembers are applied to the following items. The sum of the points received from all the questions will be divided by the total number of questions and the total score will be obtained. A high score indicates that the quality of life is increasing, a low score indicates that it is decreasing.

CONTACTS AND LOCATIONS:
Overall Officials: Berk NIMETOGLU, Medical Doctor, Study Chair — Istanbul University Faculty of Medicine Department of Orthopedics and Traumatology
Locations (1):
- Istanbul University Faculty of Medicine Department of Orthopedics and Traumatology, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
it has been stated that it is necessary to protect the patient information contained in the patient rights regulation, and since the data must be stored, no sharing will be made. If necessary, the data will be shared collectively. Data will not be shared individually.

REFERENCES:
- [Background] Hawes MC. The use of exercises in the treatment of scoliosis: an evidence-based critical review of the literature. Pediatr Rehabil. 2003 Jul-Dec;6(3-4):171-82. doi: 10.1080/0963828032000159202. PMID 14713583
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Dahl-Popolizio S, Loman J, Cordes CC. Comparing Outcomes of Kinect Videogame-Based Occupational/Physical Therapy Versus Usual Care. Games Health J. 2014 Jun;3(3):157-61. doi: 10.1089/g4h.2014.0002. Epub 2014 Apr 17. PMID 26196174